CLINICAL TRIAL: NCT02341495
Title: A Phase II Study Examining the Use of Deferasirox, Cholecalciferol, and Azacitidine in the Treatment of Newly Diagnosed Acute Myelogenous Leukemia (AML) in Elderly Patients
Brief Title: Deferasirox, Cholecalciferol, and Azacitidine in the Treatment of Newly Diagnosed AML Patients Over 65
Acronym: EXJADE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early due to low patient accrual.
Sponsor: Elizabeth Henry (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Henry, Faculty, Loyola University
Organization: Loyola University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 204961
Record Dates: First submitted 2013-09-26; First posted 2015-01-19 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Azacitidine; Vidaza; Deferasirox; Exjade; Cholecalciferol; Vitamin D
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Deferasirox; Cholecalciferol; Vitamin D; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug Treatment (Experimental): Deferasirox (20mg/kg/day)on days 1-7 of protocol, repeated every four weeks for 8 cycles given PO Cholecalciferol(4,000 units/day), on days 1-7 of protocol, repeated every four weeks for 8 cycles given PO Azacitidine (75mg/m2 subcutaneous or IV administration) on days 1-7 of protocol, repeated every four weeks for 8 cycles given either subcutaneously or IV
  Interventions: Drug: Deferasirox; Drug: Cholecalciferol; Drug: Azacitidine

INTERVENTIONS:
Drug: Deferasirox — Deferasirox (20mg/kg/day)on days 1-7 of protocol every 4 wks for 8 cycles PO
  Other Names: Exjade
Drug: Cholecalciferol — Cholecalciferol(4,000 units/day) on days 1-7 of protocol every 4 wks for 8 cycles PO
  Other Names: Vitamin D
Drug: Azacitidine — Azacitidine (75mg/m2 subcutaneous or IV administration) on days 1-7 of protocol 28 days for 32 wks
  Other Names: Vidaza

SUMMARY:
The purpose of this study is to find out if by giving a combination of 3 drugs the leukemia will go into complete remission (meaning the leukemia is completely gone), and to find out how long it stays away. The drugs used in this project are FDA approved and commercially available.

DETAILED DESCRIPTION:
The majority of new cases of acute myeloid leukemia (AML) are diagnosed in patients older than 65 years of age. The median age of patients at time of diagnosis is 67 years. Standard therapies for AML often have significant toxicity and are poorly tolerated by this patient population. Treatment strategies for elderly patients with AML are limited. In those patients who do achieve complete remission, duration of remission tends to be short. Treatment at time of relapse is exceedingly difficult and outcomes are dismal. Thus, there is need for safer and more effective therapies for elderly patients with AML. This trial is a novel therapeutic combination of deferasirox (Exjade), cholecalciferol, and azacitidine in patients 65 years or older with newly diagnosed AML who are not fit for standard induction chemotherapy or hematopoietic stem-cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 65 or older (must have reached 65th birthday)
* Morphologically confirmed diagnosis of AML, excluding AML-M3
* Must have a Zubrod performance status of 0-3

Exclusion Criteria:

* Patients with known HIV infection are excluded. If HIV infection is suspected based on clinical condition, testing may be performed at the discretion of treatment team, but is not mandated prior to enrollment.
* Patients with central nervous system involvement by AML are excluded
* Patients with history of an active cancer (except basal cell and squamous cell cancers of the skin) within the previous 2 years are excluded

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Henry, MD, Principal Investigator — Faculty
Locations (1):
- Loyola University Cardinal Bernardin Cancer Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individuals participant data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug Treatment
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Drug Treatment
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate
Description: The Complete Remission Rate for all evaluable patients will be reported for the following treatment: azacitadine, vitamin D, and deferasirox (Exjade). The proportion of patients experiencing per-protocol CR will be calculated with a 90% exact confidence interval.
Time Frame: up to 5 years
Population: No patients were analyzed as study was terminated early due to low accrual. Therefore, data necessary for planned analyses were not collected.
Arm/Group | Drug Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Patients With Adverse Events
Description: Characterization of the safety of an induction regimen of azacitidine in combination with vitamin D and deferasirox (Exjade). The proportion of patients experiencing severe adverse events, and the number of patients experiencing severe adverse events probably or definitely related to treatment will be determined. Adverse events will be tabulated by category and graded by NCI CTCAE version 4.0
Time Frame: up to 5 years
Population: as for outcome 1
Arm/Group | Drug Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Survival
Description: The overall survival and relapse-free survival functions. Product-limit (Kaplan-Meier) estimate of the survival functions will be estimated, with 90% confidence intervals.
Time Frame: up to 5 years
Population: as for outcome 1
Arm/Group | Drug Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Remission
Description: The length of time for remission after achieving complete remission
Time Frame: up to 5 years
Population: as for outcome 1
Arm/Group | Drug Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 45 months
Arm/Group | Drug Treatment
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report as the study was terminated early due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes